CLINICAL TRIAL: NCT04244786
Title: Treating Self Injurious Behavior: A Novel Brain Stimulation Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Jeffrey Miller, Associate Professor of Clinical Psychiatry, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: #7170
Record Dates: First submitted 2019-10-23; First posted 2020-01-28 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Self-Injurious Behavior; Self Harm; Self-injury; Self-inflicted Injury; Self Injurious Behavior Without Suicidal Intent; Non-Suicidal Self Injury; Non Suicidal Self Inflicted Injury; Cutting; Depression; Bipolar Disorder; Borderline Personality Disorder
Keywords: Transcranial direct current stimulation; Transcranial electric stimulation; non-invasive brain stimulation; tDCS
MeSH Terms: conditions — Self-Injurious Behavior; Depression; Bipolar Disorder; Borderline Personality Disorder | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, sham-controlled trial. 2 arms of clinical trial. Listing 3 arms to include an arm for individuals who signed consent but discontinued prior to randomization and clinical intervention, to describe available data and adverse events in this group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: tDCS device programmed with codes to deliver active vs. sham tDCS in a blinded manner. Individual independent of study team managed randomization and provided codes for blinded tDCS administration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- active anodal tDCS to ventrolateral prefrontal cortex (VLPFC) (Active Comparator): active anodal tDCS to ventrolateral prefrontal cortex (VLPFC).
  1.5 milliamp (mA) anodal tDCS over right ventrolateral prefrontal cortex; 12 20-minute administrations over 6-sessions
  Interventions: Device: Transcranial direct current stimulation
- sham anodal tDCS to VLPFC (Sham Comparator): sham anodal tDCS to VLPFC
  Identical electrode montage, 12 administrations of sham tDCS over 6 sessions.
  Interventions: Device: Transcranial direct current stimulation
- Discontinued prior to randomization (Other): Participants who enrolled in the study but discontinued before being randomized to either active or sham arms of the study
  Interventions: Other: No intervention

INTERVENTIONS:
Device: Transcranial direct current stimulation — tDCS is a low-cost, portable, well-tolerated, non-invasive form of brain stimulation that delivers a low current to a specific area of the brain via electrodes.
  Arms: active anodal tDCS to ventrolateral prefrontal cortex (VLPFC); sham anodal tDCS to VLPFC
Other: No intervention — No intervention for participants who discontinued prior to randomization
  Arms: Discontinued prior to randomization

SUMMARY:
The purpose of this study is to explore the tolerability and effectiveness of transcranial direct current stimulation (tDCS) as a potential treatment for non-suicidal self-injury (NSSI). Individuals who engage in frequent NSSI will be randomized to 12 administrations of an active vs. inactive form of tDCS, paired with an Attention Training Technique task, over a two-week period. Functional MRI may be performed before and after this two week period. NSSI urges and behaviors will be monitored before, during, and after the period of tDCS administrations.

DETAILED DESCRIPTION:
The purpose of this study is to explore the tolerability and effectiveness of transcranial direct current stimulation (tDCS) as a potential treatment for non-suicidal self-injury (NSSI). NSSI is the deliberate attempt to harm oneself, most often through cutting or burning, without suicidal intent. NSSI is a maladaptive emotion-regulation strategy often triggered by negative emotions, especially those involving feelings of rejection. tDCS is a low-cost, portable, well-tolerated, non-invasive form of brain stimulation that delivers a low current to a specific area of the brain via electrodes. Several studies have demonstrated its effectiveness in treating an array of conditions, depending on electrode placement, including depression and chronic pain. tDCS may also facilitate adaptive emotion regulation; researchers have also successfully used tDCS to reduce negative emotions and aggressive responses to social rejection. The investigators therefore seek to explore tDCS as a potential treatment for NSSI. This pilot feasibility study seeks 1) to examine how tDCS is tolerated in a sample of individuals who engage in frequent NSSI; 2) to gather pilot data regarding changes in emotional and neural responses during a social task after a series of tDCS sessions in this clinical population of individuals who engage in NSSI; 3) to gather pilot data on the effects of tDCS on NSSI behaviors and urges. The investigators seek to recruit a sample of 22 individuals who engage in frequent NSSI to complete all study procedures. Individuals will be randomized to receive active- or sham-tDCS for two twenty-minute applications on each of six alternating sessions over approximately two weeks for a total of 12 tDCS administrations, each paired with an Attention Training Task. Functional MRI (fMRI) may be performed at baseline and again after the completion of 12 applications of tDCS. Subjects' NSSI and urges to engage in NSSI will be recorded for four weeks in real-time, using an iPod- based system that reminds subjects to stop at certain times during the day to record their thoughts, feelings, and behaviors. This will allow measurement of NSSI urges and behaviors for one week before, two weeks during, and one week after the tDCS intervention. The long-term goal of this study is to identify a novel form of treatment for NSSI and to better understand NSSI pathophysiology.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60
2. Frequent current NSSI (including cutting in which the skin is broken; self-hitting in which there is bruising; or burning in which there is evidence of a burn. Will not enroll if skin-picking or scratching is the only form of self-injury): has engaged in ≥2 episodes of NSSI in the two months prior to enrollment
3. Capacity to provide informed consent
4. If carries a diagnosis of bipolar I or II disorder, taking or willing to begin a therapeutic dose of a mood stabilizer.
5. Normal hearing.
6. Physical capacity (e.g., manual dexterity) to set-up and self-administer tDCS. -

Exclusion Criteria:

1. Unstable medical conditions based on medical history or physical examination
2. Current psychotic disorder, mania, hypomania, intellectual disability
3. Dermatologic condition resulting in non-intact skin on the scalp
4. Significant suicidal ideation with a plan and intent that cannot be managed safely as an outpatient
5. Pregnancy, currently lactating, or planning to conceive during the course of study participation.
6. A neurological disease or prior head trauma with evidence of cognitive impairment. Subjects who endorse a history of prior head trauma and score ≥ 1.5 standard deviations below the mean on the Trailmaking A&B will be excluded from study participation.
7. Current alcohol or substance use disorder that is severe according to DSM-V criteria
8. Individuals who initiated or increased the dose of concurrent psychiatric medications (including antidepressants, anxiolytics, antipsychotic medications, mood stabilizers, and benzodiazepines) within two weeks prior to enrollment
9. Individuals who initiated psychotherapy within two weeks prior to enrollment
10. Current seizure disorder.
11. Use of anticonvulsant medications that target the GABA system (e.g., gabapentin).
12. Individuals currently using benzodiazepines who are unwilling or unable to refrain from the use of benzodiazepine medications for at least 72 hours before the first tDCS session and throughout the duration of the 2-week tDCS intervention.
13. Metal implants or paramagnetic objects contained within the body (including heart pacemaker, shrapnel, or surgical prostheses) which may present a risk to the subject or interfere with the MRI scan, according to the guidelines set forth in the following reference book commonly used by neuroradiologists: "Guide to MR procedures and metallic objects," F.G. Shellock, Lippincott Williams and Wilkins NY 2001. Additionally transdermal patches will be removed during the MR study at the discretion of the investigator.
14. Claustrophobia significant enough to interfere with MRI scanning
15. Weight that exceeds 325 lbs or inability to fit into MRI scanner
16. Suicide attempt within the past 3 months
17. Serious self-harm resulting in hospitalization within the past 3 months.

    -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M Miller, MD, Principal Investigator — NYSPI
Locations (1):
- New York State Psychiatric Institute/Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Scan results, questionnaire answers, and data collected during the task may be used in future studies, and if shared with other investigators, information that identifies the scan, questionnaire responses, or task data with you will be removed before hand.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: upon request
Access Criteria: upon request

REFERENCES:
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Anodal tDCS to Ventrolateral Prefrontal Cortex (VLPFC): active anodal tDCS to ventrolateral prefrontal cortex (VLPFC).
  1.5 milliamp (mA) anodal tDCS over right ventrolateral prefrontal cortex; 12 20-minute administrations over 6-sessions
  Transcranial direct current stimulation: tDCS is a low-cost, portable, well-tolerated, non-invasive form of brain stimulation that delivers a low current to a specific area of the brain via electrodes.
- Sham Anodal tDCS to VLPFC: sham anodal tDCS to VLPFC
  Identical electrode montage, 12 administrations of sham tDCS over 6 sessions.
  Transcranial direct current stimulation: tDCS is a low-cost, portable, well-tolerated, non-invasive form of brain stimulation that delivers a low current to a specific area of the brain via electrodes.
Period: Overall Study
Arm/Group | Active Anodal tDCS to Ventrolateral Prefrontal Cortex (VLPFC) | Sham Anodal tDCS to VLPFC | Discontinued Prior to Randomization
Started | 3 | 3 | 7
Completed | 3 | 3 | 0
Not Completed | 0 | 0 | 7
Not completed — Adverse Event | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 5

BASELINE CHARACTERISTICS:
Population: Participants with non-suicidal self-injurious behavior (at least 2 episodes in the past 2 months) who met study criteria and consented to the study protocol.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Anodal tDCS to Ventrolateral Prefrontal Cortex (VLPFC) | Sham Anodal tDCS to VLPFC | Discontinued Prior to Randomization | Total
Number analyzed (Participants) | 3 | 3 | 7 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.7 (3.5) | 20 (1) | 25.1 (6.0) | 23.8 (5.0)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Self-reported gender identity
  Participants
    Female | 3 | 2 | 5 | 10
    Male | 0 | 0 | 1 | 1
    Non-Binary | 0 | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 2
  Not Hispanic or Latino | 3 | 3 | 5 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 2 | 2 | 6 | 10
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Social Processing (Cyberball) fMRI Task: fMRI Responses
Description: The Cyberball task is a task used during functional MRI scanning. During the task, individuals play a virtual ball-tossing game, playing catch with two computer avatars, and have a social exclusion experience when the avatars stop tossing the ball to them. The outcome measure is a subtraction of a measure of brain activity (fMRI BOLD signal) during portions of the task when the individual is included in the virtual ball-tossing game as compared to periods when the individual is excluded (i.e. fMRI BOLD signal inclusion periods - fMRI BOLD signal exclusion periods). This is quantified in 7 specific brain regions specified in the table below. dACC = dorsal anterior cingulate. vlPFC = ventrolateral prefrontal cortex. AI = anterior insula. The unit of measurement is a beta-weight from a general linear model (a statistical model) and a higher value reflects greater activity in a given brain region during experiences of social exclusion as compared to social inclusion.
Time Frame: Pre-treatment (baseline) and post-treatment (up to 2 weeks)
Measure: Mean (Standard Deviation); unit: beta-weight
Groups:
- Sham Anodal tDCS to VLPFC: Pre-treatment; Sham Anodal tDCS to VLPFC: Post-treatment: Identical electrode montage, 12 administrations of sham tDCS over 6 sessions.
- Active Anodal tDCS to Ventrolateral Prefrontal Cortex (VLPFC): Pre-treatment: 1.5 milliamp (mA) anodal tDCS over right ventrolateral prefrontal cortex; 12 20-minute administrations over 6-sessions
- Active Anodal tDCS to Ventrolateral Prefrontal Cortex (VLPFC): Post-treatment: 1.5 milliamp (mA) anodal tDCS over right ventrolateral prefrontal cortex; 12 20-minute administrations over 6 sessions
Arm/Group | Sham Anodal tDCS to VLPFC: Pre-treatment | Sham Anodal tDCS to VLPFC: Post-treatment | Active Anodal tDCS to Ventrolateral Prefrontal Cortex (VLPFC): Pre-treatment | Active Anodal tDCS to Ventrolateral Prefrontal Cortex (VLPFC): Post-treatment | Discontinued Prior to Randomization
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2
beta-weight
  Parcel 29 (left dACC) | -621.4739585 (819.58606846675) | -519.1597701 (1187.3713291081) | -63.33972338 (851.26348872338) | -396.4460666 (779.73833545212) | 286.13477133333 (1560.1228270282)
  Parcel 183 (right dACC) | -651.4402542 (1422.0518670889) | -581.3360775 (1419.4881641560) | -324.0953143 (1101.3079494312) | -168.76175 (679.73029181028) | 384.62016755555 (2082.2972871030)
  Parcel 240 (right vlPFC) | -227.9885197 (395.65696014195) | -203.971185 (671.54324931238) | 446.1573213 (650.27267162975) | -287.2243125 (839.18680962738) | -588.4478376 (1036.4740809912)
  Parcel 241 (right vlPFC) | -335.4290303 (565.88946960588) | -215.3886576 (1194.5755014134) | 50.34725113 (456.40817606524) | 57.968314699999 (956.33384050042) | -482.2452623 (1373.3034293132)
  Parcel 242 (right vlPFC) | -756.0566932 (956.69043909054) | -297.5780364 (1289.3740570339) | 320.32500074999 (986.09839303323) | 48.925466799999 (730.94081312280) | -264.4217283 (1149.8191589249)
  Parcel 247 (right AI) | -247.2044975 (466.61315305963) | -495.6796714 (758.72874358403) | -127.9602427 (1163.6302170131) | -93.3563077 (888.06111718986) | -141.689008 (1181.0573804472)
  Parcel 281 (right vlPFC) | -234.9502234 (454.57709537062) | -229.4499879 (706.92156796310) | 220.64673762500 (609.39673885219) | -137.8113024 (437.9420888) | -179.9291584 (1004.2419972306)

2. Primary Outcome: Ecological Momentary Assessment (EMA): Duration, Intensity, and Severity of NSSI Urges and Behavior
Description: EMA assessment of NSSI urges and behavior before, during, and after tDCS intervention. EMA is a tool through which participants can respond to a brief questionnaire on a smartphone device while going about their daily lives. Participants were prompted to complete a brief questionnaire 6 times per day over a 4 week period (one week before tDCS (baseline), 2 weeks during tDCS (during tDCS), and one week after the final tDCS administration (post-tDCS)), which asks questions about urges to engage in NSSI and in actual NSSI behavior. Scores, coded on a scale from 1-5, are averaged across all prompts during the time period (baseline, during tDCS, post-tDCS). A higher score indicates more severe symptoms except for "success at resisting thoughts", which is reverse-coded.
Time Frame: One week before tDCS (baseline), two weeks during tDCS (during tDCS), one week post-tDCS (post-tDCS)
Measure: Mean (Standard Deviation); unit: Average score on a scale
Groups:
- Sham Anodal tDCS to Ventrolateral Prefrontal Cortex (VLPFC): Identical electrode montage, 12 administrations of sham tDCS over 6 sessions.
- Active Anodal tDCS to VLPFC: 1.5 milliamp (mA) anodal tDCS over right ventrolateral prefrontal cortex; 12 20-minute administrations over 6-sessions
Arm/Group | Sham Anodal tDCS to Ventrolateral Prefrontal Cortex (VLPFC) | Active Anodal tDCS to VLPFC
Number analyzed (Participants) | 3 | 3
Average score on a scale
  Strength of self-injury thoughts: baseline | 1.2697 (0.6952) | 1.5285 (1.0736)
  Strength of self-injury thoughts: during tDCS | 1.1186 (0.7094) | 1.2294 (0.9414)
  Strength of self-injury thoughts: post-tDCS | 0.5667 (0.8014) | 1.38 (0.9439)
  Duration of self-injury thoughts: baseline | 0.9821 (0.4538) | 1.2479 (1.1492)
  Duration of self-injury thoughts: during tDCS | 0.6770 (0.3366) | 0.9503 (0.9765)
  Duration of self-injury thoughts: post-tDCS | 0.3333 (0.4714) | 1.2307 (0.9196)
  Difficulty resisting self-injury thoughts: baseline | 1.0587 (0.6349) | 1.0711 (0.8945)
  Difficulty resisting self-injury thoughts: during tDCS | 1.0636 (0.8165) | 0.9338 (0.93)
  Difficulty resisting self-injury thoughts: post-tDCS | 0.5667 (0.8014) | 0.7879 (1.0654)
  Success at resisting self-injury thoughts: baseline | 1.0774 (0.8346) | 0.8344 (0.5786)
  Success at resisting self-injury thoughts: during tDCS | 1.0476 (0.8987) | 0.7404 (0.6601)
  Success at resisting self-injury thoughts: post-tDCS | 0.6667 (0.9428) | 0.4444 (0.5092)

3. Primary Outcome: Self Injurious Thoughts and Behaviors Inventory Part 1
Description: Selected items from the Self-Injurious Thoughts and Behaviors Interview (SITBI) were used at baseline and after the tDCS or sham intervention as outcome measures in this study. These items ask participants to report on their NSSI thoughts and behaviors over the past week. The following items are reported in this table:
  Sitbi 58: At their worst, how intense were your thoughts about engaging in NSSI? (0: very mild to 4: very severe) sitbi 59: On average, how intense were your thoughts about engaging in NSSI? (0: very mild to 4: very severe)
Time Frame: Pre-treatment (baseline) and post-tDCS (up to 2 weeks after baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Sham Anodal tDCS to VLPFC: Baseline; Sham Anodal tDCS to VLPFC: Post tDCS: Identical electrode montage, 12 administrations of sham tDCS over 6 sessions
- Active Anodal tDCS to Ventrolateral Prefrontal Cortex (VLPFC): Baseline; Active Anodal tDCS to Ventrolateral Prefrontal Cortex (VLPFC): Post-tDCS: 1.5 milliamp (mA) anodal tDCS over right ventrolateral prefrontal cortex; 12 20-minute administrations over 6-sessions
Arm/Group | Sham Anodal tDCS to VLPFC: Baseline | Sham Anodal tDCS to VLPFC: Post tDCS | Active Anodal tDCS to Ventrolateral Prefrontal Cortex (VLPFC): Baseline | Active Anodal tDCS to Ventrolateral Prefrontal Cortex (VLPFC): Post-tDCS
Number analyzed (Participants) | 3 | 3 | 3 | 3
score on a scale
  At their worst, how intense were your thoughts about engaging in self-harm? (sitbi 58) | 2.33 (1.15) | 2.67 (1.15) | 2.67 (0.58) | 2.67 (1.15)
  On average, how intense were your thoughts about engaging in self-harm? (sitbi 59) | 1.67 (0.58) | 2 (1) | 1.67 (0.58) | 2.33 (0.58)

4. Primary Outcome: Ecological Momentary Assessment (EMA): NSSI Urges and Behavior
Description: EMA assessment of NSSI urges and behavior before, during, and after tDCS intervention. EMA is a tool through which participants can respond to a brief questionnaire on a smartphone device while going about their daily lives. Participants were prompted to complete a brief questionnaire 6 times per day over a 4 week period (one week before tDCS (baseline), 2 weeks during tDCS (during tDCS), and one week after the final tDCS administration (post-tDCS)), which asks questions about urges to engage in NSSI and in actual NSSI behavior. Items refer to the proportion of survey responses in which an individual endorsed the given thought or behavior or attempted to resist NSSI thoughts since the previous response (0 to 1), with "yes" scored as 1 and "no" scored as a zero.
Time Frame: One week before tDCS (baseline), two weeks during tDCS (during tDCS), one week post-tDCS (post-tDCS)
Measure: Mean (Standard Deviation); unit: Proportion of prompts
Arm/Group | Sham Anodal tDCS to Ventrolateral Prefrontal Cortex (VLPFC) | Active Anodal tDCS to VLPFC
Number analyzed (Participants) | 3 | 3
Proportion of prompts
  Thoughts of self-injury: baseline | 0.4453 (0.2874) | 0.4664 (0.2274)
  Thoughts of self-injury: during tDCS | 0.4084 (0.2963) | 0.3661 (0.2166)
  Thoughts of self-injury: post-tDCS | 0.2333 (0.33) | 0.3937 (0.2379)
  Attempted to resist self-injury thoughts: baseline | 0.3658 (0.2531) | 0.3146 (0.2470)
  Attempted to resist self-injury thoughts: during tDCS | 0.3509 (0.2937) | 0.2803 (0.2644)
  Attempted to resist self-injury thoughts: post-tDCS | 0.2 (0.2828) | 0.2071 (0.2608)
  Self-harm behavior: baseline | 0.0975 (0.1082) | 0.1759 (0.1818)
  Self-harm behavior: during tDCS | 0.1261 (0.1615) | 0.1073 (0.1298)
  Self-harm behavior: post-tDCS | 0.1 (0.1414) | 0.0967 (0.1343)

5. Primary Outcome: Self Injurious Thoughts and Behaviors Inventory Part 2
Description: Selected items from the Self-Injurious Thoughts and Behaviors Interview (SITBI) were used at baseline and after the tDCS or sham intervention as outcome measures in this study. These items ask participants to report on their NSSI thoughts and behaviors over the past week. The following item is reported in this table:
  sitbi 68: How many times [did you self-injure] in the past week? (number entered, minimum = 0, maximum = no limit)
Time Frame: pre-treatment (baseline) and post-treatment (up to 2 weeks)
Measure: Mean (Standard Deviation); unit: Number of events
Arm/Group | Sham Anodal tDCS to VLPFC: Baseline | Sham Anodal tDCS to VLPFC: Post tDCS | Active Anodal tDCS to Ventrolateral Prefrontal Cortex (VLPFC): Baseline | Active Anodal tDCS to Ventrolateral Prefrontal Cortex (VLPFC): Post-tDCS
Number analyzed (Participants) | 3 | 3 | 3 | 3
Number of events | 4.33 (2.52) | 1.33 (0.58) | 9.67 (13.43) | 1.33 (2.31)

6. Primary Outcome: Self Injurious Thoughts and Behaviors Inventory Part 3
Description: Selected items from the Self-Injurious Thoughts and Behaviors Interview (SITBI) were used at baseline and after the tDCS or sham intervention as outcome measures in this study. These items ask participants to report on their NSSI thoughts and behaviors over the past week. The following item is reported in this table:
  sitbi 60: When you have had these thoughts: how long have they usually lasted? (0: 0 seconds to 6: more than 2 days)
Time Frame: Pre-treatment (baseline) and post-tDCS (up to 2 weeks after baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham Anodal tDCS to VLPFC: Baseline | Sham Anodal tDCS to VLPFC: Post tDCS | Active Anodal tDCS to Ventrolateral Prefrontal Cortex (VLPFC): Baseline | Active Anodal tDCS to Ventrolateral Prefrontal Cortex (VLPFC): Post-tDCS
Number analyzed (Participants) | 3 | 3 | 3 | 3
score on a scale | 2.33 (0.58) | 2.33 (1.15) | 3.33 (0.58) | 3.33 (2.31)

7. Primary Outcome: Self Injurious Thoughts and Behaviors Inventory Part 4
Description: Selected items from the Self-Injurious Thoughts and Behaviors Interview (SITBI) were used at baseline and after the tDCS or sham intervention as outcome measures in this study. These items ask participants to report on their NSSI thoughts and behaviors over the past week. The following items are reported here:
  sitbi 61: What is the likelihood you will have thoughts about engaging in NSSI in the future? (0: very unlikely to 4: very likely) sitbi 72: What do you think is the likelihood you will engage in NSSI in the future? (0: very unlikely to 4: very likely)
Time Frame: Pre-treatment (baseline) and post-tDCS (up to 2 weeks after baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham Anodal tDCS to VLPFC: Baseline | Sham Anodal tDCS to VLPFC: Post tDCS | Active Anodal tDCS to Ventrolateral Prefrontal Cortex (VLPFC): Baseline | Active Anodal tDCS to Ventrolateral Prefrontal Cortex (VLPFC): Post-tDCS
Number analyzed (Participants) | 3 | 3 | 3 | 3
score on a scale
  Likelihood of future self-harm thoughts (sitbi 61) | 4 (0) | 33 (0.58) | 4 (0) | 4 (0)
  Likelihood of future self-harm (sitbi 72) | 4 (0) | 3.33 (0.58) | 3.67 (0.58) | 3.67 (0.58)

8. Other Pre Specified Outcome: tDCS Adverse Effects Questionnaire
Description: A questionnaire to evaluate side-effects related to tDCS administration. This questionnaire asks about the presence and severity of possible side-effects of tDCS procedures, and was recently published as a gold-standard tool for this purpose: Aparício LVM, Guarienti F, Razza LB, Carvalho AF, Fregni F, Brunoni AR. A Systematic Review on the Acceptability and Tolerability of Transcranial Direct Current Stimulation Treatment in Neuropsychiatry Trials. Brain Stimul. 2016 Oct;9(5):671-81. This is an 11-item scale, that asks about the occurrence and severity of a range of possible side-effects during or after tDCS administration. Each side-effect can be rated as absent, mild, moderate, or severe. Summary data regarding the number of participants who endorsed a listed side-effect from the scale during at least one tDCS administration are presented here. Each participant was asked about the presence and severity of all listed side-effects after each administration of tDCS.
Time Frame: Administered after each (12) tDCS session over 6 days
Measure: Count of Participants; unit: Participants
Groups:
- Sham Anodal tDCS to VLPFC: Identical electrode montage, 12 administrations of sham tDCS over 6 sessions.
- Active Anodal tDCS to Ventrolateral Prefrontal Cortex (VLPFC): 1.5 milliamp (mA) anodal tDCS over right ventrolateral prefrontal cortex; 12 20-minute administrations over 6-sessions
Arm/Group | Sham Anodal tDCS to VLPFC | Active Anodal tDCS to Ventrolateral Prefrontal Cortex (VLPFC)
Number analyzed (Participants) | 3 | 3
Participants
  Headache | 2 | 2
  Neck Pain | 0 | 1
  Scalp pain | 1 | 1
  Tingling | 3 | 2
  Itching | 3 | 2
  Burning sensation | 3 | 3
  Skin Redness | 3 | 3
  Sleepiness | 3 | 2
  Trouble concentrating | 3 | 3
  Acute mood change | 0 | 3
  Other | 1 | 2

ADVERSE EVENTS:
Time Frame: For study completers: >4 weeks. Study procedures occur over an approx 4 week period (1 week prior to tDCS procedures, 2 weeks of tDCS procedures, 1 week following tDCS procedures). However, there is generally some time from signing of consent to scheduling of baseline research procedures. In general, time frame is approximately 7-8 weeks for study completers. For individuals who discontinued prior to randomization, time frame is from consent to study discontinuation, generally 1 to 3 weeks.
Description: Possible side-effects during tDCS administration were assessed using a structured instrument, the tDCS Adverse Effects Questionnaire, administered after each tDCS administration. While not all physical experiences endorsed on the scale represent an adverse event, all endorsements from the scale are reported here for thoroughness.
Groups:
- Sham Anodal tDCS to Ventrolateral Prefrontal Cortex (VLPFC): Identical electrode montage, 12 administrations of sham tDCS over 6 sessions.
  Transcranial direct current stimulation: tDCS is a low-cost, portable, well-tolerated, non-invasive form of brain stimulation that delivers a low current to a specific area of the brain via electrodes.
Arm/Group | Sham Anodal tDCS to Ventrolateral Prefrontal Cortex (VLPFC) | Active Anodal tDCS to Ventrolateral Prefrontal Cortex (VLPFC) | Discontinued Prior to Randomization
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 2/7
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham Anodal tDCS to Ventrolateral Prefrontal Cortex (VLPFC) (N=3) | Active Anodal tDCS to Ventrolateral Prefrontal Cortex (VLPFC) (N=3) | Discontinued Prior to Randomization (N=7)
Hospitalization (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Medical hospitalization for non-suicidal self-injury that occurred one day after consent, prior to any research procedures beyond evaluation and consent, unrelated to research participation.
Suicide Attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) — Individual crossed the street without looking, indifferent to outcome. No medical injury. Individual did not consider this a suicide attempt, but was categorized as such by our research classification. Occurred prior to randomization.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham Anodal tDCS to Ventrolateral Prefrontal Cortex (VLPFC) (N=3) | Active Anodal tDCS to Ventrolateral Prefrontal Cortex (VLPFC) (N=3) | Discontinued Prior to Randomization (N=7)
Headache (Nervous system disorders) | 2 (13) | 2 (15) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Scalp Pain (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Tingling (Skin and subcutaneous tissue disorders) | 3 (12) | 2 (15) | 0 (0)
Itching (Skin and subcutaneous tissue disorders) | 3 (17) | 2 (16) | 0 (0)
Burning Sensation (Skin and subcutaneous tissue disorders) | 3 (26) | 3 (32) | 0 (0)
Skin redness (Skin and subcutaneous tissue disorders) | 3 (35) | 3 (31) | 0 (0)
Sleepiness (Nervous system disorders) | 3 (25) | 2 (15) | 0 (0)
Trouble concentrating (Nervous system disorders) | 3 (25) | 3 (29) | 0 (0)
Acute Mood Change (Psychiatric disorders) | 0 (0) | 3 (4) | 0 (0)
Other: Heart palpitations (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0)
Other: Psychomotor agitation (Psychiatric disorders) | 0 (0) | 1 (3) | 0 (0) — Symptom write-in for "other" option. Participant reported feeling "fidgety"
Other: Derealization (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) — Participant wrote in "spacey feeling" for "other" selection
Other: Pressure (Product Issues) | 1 (1) | 0 (0) | 0 (0) — Participant reported uncomfortable tightness from the headstrap

LIMITATIONS AND CAVEATS:
Small sample size recruited allow for analyses for hypothesis generation and preliminary data supporting future, larger studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-29): https://cdn.clinicaltrials.gov/large-docs/86/NCT04244786/Prot_SAP_000.pdf